CLINICAL TRIAL: NCT02661698
Title: Diurnal Variation of Plasma Concentration of EPA and DHA and Absorption of Doses Taken at Hora Somni
Brief Title: Plasma Diurnal Variation in and Absorption of EPA and DHA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northumbria University (Other)
Collaborators: Pronova BioPharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple
Other Study IDs: 44N2
Record Dates: First submitted 2016-01-14; First posted 2016-01-22 (Estimated); Last update posted 2016-11-08 (Estimated); Status verified 2016-09

CONDITIONS: Lipid Absorption and Metabolism

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Placebo 1 (Placebo Comparator): Placebo
  All participants will be given a placebo for the first visit. The other 3 arms will be randomised in a counterbalanced order.
  Interventions: Dietary Supplement: Placebo
- Placebo 2 (Placebo Comparator): Placebo
  Interventions: Dietary Supplement: Placebo
- DHA rich oil (Active Comparator): Omega-3 oil: DHA enriched
  Interventions: Dietary Supplement: Omega-3 oil: DHA enriched
- EPA rich oil (Active Comparator): Omega-3 oil: EPA enriched
  Interventions: Dietary Supplement: Omega-3 oil: EPA enriched

INTERVENTIONS:
Dietary Supplement: Omega-3 oil: DHA enriched — 3 x 1 g capsules containing a SMEDDS formulation of an DHA-enriched oil: 50% DHA + 15% EPA totalling 900 mg DHA and 270 mg of EPA
  Arms: DHA rich oil
Dietary Supplement: Placebo — 3 x 1 g capsules Placebo: olive oil
  Arms: Placebo 1; Placebo 2
Dietary Supplement: Omega-3 oil: EPA enriched — 3 x 1 g capsules containing a SMEDDS formulation of an EPA-enriched oil: 50% EPA + 20% DHA totalling 900 mg EPA and 360 mg of DHA
  Arms: EPA rich oil

SUMMARY:
This study will evaluate the absorption of two different dietary supplements containing the omega 3 fatty acids eicosapentaenoic acid and docosahexaenoic acid over 24 hours via venous blood plasma following a single dose taken at bed time. In addition, the circadian rhythm of fatty acid metabolism will also be assessed following the placebo intervention.

DETAILED DESCRIPTION:
The bioavailability of the omega-3 fatty acids eicosapentaenoic acid (EPA) and docosahexaenoic acid (DHA) can be influenced by a number of factors including chemical structure of the fatty acid binding form and the food matrix with which the fatty acids are consumed. In addition to this, there is evidence from animals that the lipid metabolism follows a circadian pattern, although this has yet to be investigated in humans.

The supplement is produced as a soft gelatine capsule containing fish oil based high concentrate omega-3 fatty acids designed to improve bio availability via a self-emulsifying drug delivery system (SMEDDS). The in-situ formation of an emulsion occurs spontaneously when the capsule erupts in vivo and the SMEDDS solution comes in contact with the gastro-intestinal contents. The size of the microdroplets that are formed is in the lower micrometer range, the advantage of which is a much larger combined surface area compared to drops of oil which results in better access for pancreatic lipases. The resulting free fatty acids may then readily be absorbed during its passage through the upper small intestine resulting in an effective absorption of the oil.

Therefore duel objectives of this study are to determine the bioavailability in healthy middle aged adults of two formulations of fish oil taken at bed time using SMEDDS and to evaluate the diurnal variation in background plasma fatty acids.

All study visits will take place on the 4th floor of the Northumberland Building, Northumbria University within a suite of facilities comprising the Nutrition Kitchen, Sleep Centre, Clinical space and the waiting room of the Brain, Performance and Nutrition Research Centre. Participants will attend the lab on five separate occasions. The first visit will be a screening/introductory visit. The Introductory visit to the laboratory will comprise: providing each participant with a 'participant information sheet', briefing them on the requirements of the study and signing of the informed consent form and completion of the Case Report Form (CRF; including self-reported health screening and collection of demographic data). Participants will then attend the lab for four study visits which will be separated by at least 6 days, each of which will be identical except for the treatment that they will consume. On each of the study visits participants will arrive at the lab at 19:30 having consumed nothing but water for at least 2 hours prior to their arrival where their continued eligibility will be assessed. A cannula will then be inserted into a vein in the arm of the non-dominant hand. The first blood sample will be collected immediately prior to their evening meal which will be served at 20:00 and will be followed by a rest period. At 22:00 participants will consume their evening's treatment. Lights out will be at 22:30. Blood samples will be drawn every 2 hours through the night at 00:00, 02:00 and 04:00. Participants will be woken up at 06:00 and a blood sample will be taken straight away. Blood samples will continue to be collected every two hours until 22:00 when the cannula will be removed. Meals will be provided at 07:00, 12:00, 16:00 and 20:00, with the evening meal being exactly the same as the previous evening. Participants will have ad libitum access to water throughout the study visit. They will also be allowed to consume tea and coffee throughout the day however the content and the timing of the hot drinks they consume on the first study visit will be replicated for the subsequent visits. Similarly, if they do not eat all of the meals that are provided in their entirety, this will be recorded and replicated for the subsequent visits. In between meals and blood samples participants will be required to remain within the facilities where they will be allowed to read, write, watch television or listen to music.

ELIGIBILITY:
Inclusion Criteria:

* Aged 25 to 49 years inclusive
* Males and females
* Of any ethnic origin
* Self-report of good health

Exclusion Criteria:

* • Habitual consumption of oily fish exceeds one fish meal per week

  * Consumption of omega-3 dietary supplements in the previous 4 weeks
  * Are a smoker or consume any nicotine replacement products (e.g. chewing gum, e-cigarettes)
  * Food allergies or sensitivities to any of the ingredients contained in the investigational product or any other foodstuff
  * History or current diagnosis of drug/alcohol abuse
  * Currently participating in or in the past 4 weeks participated in other clinical or nutrition intervention studies
  * High blood pressure (systolic over 159 mm Hg or diastolic over 99 mm Hg)
  * Body Mass Index outside of the range 18-35 kg/m2
  * Pregnant, trying to get pregnant or breast feeding
  * Blood donation of more than 300 mL during the three months prior to screening (470 mL is given at the average donation).
  * Sleep disturbances and/or are taking sleep aid medication
  * Currently taking blood thinning medication (e.g. aspirin, warfarin, heparin)
  * Habitually use of dietary supplements within the last month (defined as more than 3 consecutive days or 4 days in total)
  * Blood disorders (e.g. anaemia, haemophilia, thrombocytosis)
  * Diagnosis of type I or type II diabetes
  * Heart disorder, or vascular illness
  * History of kidney or liver disease, or other severe diseases of the gastrointestinal tract (e.g. iron accumulation, iron utilization disorders, hypercalcaemia, hypercalcaemia), that are likely to interfere with metabolism/absorption/secretion of the product under investigation
  * History of neurological or psychiatric illness (excluding depressive illness and anxiety)
  * Current diagnosis of depression and/or anxiety
  * Over- or under-active thyroid
  * Chronic gastrointestinal problems (e.g. Inflammatory Bowel Disease, Irritable Bowel Syndrome, celiac disease)
  * Any known active infections
  * Diagnosed with or may be at risk of having syphilis, hepatitis, the Human T - lymphotropic virus or the Human Immunodeficiency Virus?
  * Current or past breast cancer diagnosis and/or a mastectomy
  * Health condition that would prevent fulfilment of the study requirements

Ages: 25 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 39 (Actual)
Dates: Start 2016-02; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
The 24 hour Area Under the Curve (AUC) of plasma concentrations of DHA and EPA | 24 hours
  In order to assess the absorption and its effect on total exposure of each treatment in comparison to placebo, plasma data will be used to calculate the 24 hour Area Under the Curve (AUC) for the fatty acids DHA and EPA.

SECONDARY OUTCOMES:
Mesor of plasma fatty acids (DHA and EPA) | 24 hours
  The mesor is a circadian rhythm-adjusted mean based on the parameters of a cosine function fitted to the raw data
Acrophase of plasma fatty acids (DHA and EPA) | 24 hours
  the time at which the peak value is measured

CONTACTS AND LOCATIONS:
Overall Officials: Philippa A Jackson, PhD, Principal Investigator — Northumbria University
Locations (1):
- Northumbria University, Newcastle upon Tyne, Tyne and Wear, United Kingdom